CLINICAL TRIAL: NCT03988049
Title: Comparison of a 1,550 Nanometer Erbium: Glass Fractional Laser and 755-nanometer Alexandrite Picosecond Pulse Duration Laser With Diffractive Lens Array in the Treatment of Acne Scars: a Randomized, Split-face Trial
Brief Title: Comparison of 1,550 and 755 Laser in a Split-face Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: David Smart (Other)
Responsible Party: Sponsor-Investigator, David Smart, Principal Investigator, University of Utah
Organization: University of Utah (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB_00095294
Record Dates: First submitted 2017-12-06; First posted 2019-06-17 (Actual); Results first posted 2021-06-29 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Acne Scars - Mixed Atrophic and Hypertrophic
MeSH Terms: conditions — Hypertrophy

STUDY DESIGN:
Intervention Model Description: All subjects will receive half of their faces treated with each laser. Subjects will be randomized to determine which side of the face is treated with each laser.
Who Masked: Outcomes Assessor
Masking Description: Blinded Assessors will be reviewing and scoring the photos after the study is completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- 1,550 laser (Active Comparator): This arm is the side of the face treated with the 1550-nanometer Fracionated Photothermolysis laser.
  Interventions: Device: 1,550 fracionated photothermolysis laser
- 755 laser (Active Comparator): This arm is the side of the face treated with the 755-nanometer alexandrite picosecond laser.
  Interventions: Device: 755 picosecond laser

INTERVENTIONS:
Device: 1,550 fracionated photothermolysis laser — All subjects will have one side of their face treated with one laser, and the other side with the other laser.
  Arms: 1,550 laser
Device: 755 picosecond laser — All subjects will have one side of their face treated with one laser, and the other side with the other laser.
  Arms: 755 laser

SUMMARY:
Clinical Trial comparing the 1,550-nanometer fractionated photothermolysis system laser to the 755 nanometer picosecond laser using a split-face (Right-Left) comparison. Patients will receive laser treatments at week 0, week 4, and week 8. Photographs will be taken prior to laser treatment at each visit, and at the week 24 follow-up visit. Photographs will be reviewed by blinded assessors to rate each side of the face and change from baseline photos.

DETAILED DESCRIPTION:
This is a Clinical Trial comparing the 1,550-nanometer fractionated photothermolysis system laser to the 755 nanometer picosecond laser using a split-face (Right-Left) comparison. Both of these lasers are currently FDA approved for acne scarring.

Approximately 18 subjects, men and women with Fitzpatrick skin types I through V and facial acne scarring of grades III-IV (moderate to severe) will be enrolled. Both sides of the participants' face should have similar amount and severity of acne scarring. Participants will be over 18 years old. Patients have to be otherwise healthy without a history of skin cancer, keloidal scarring, localized or active infection, immunodeficiency disorders, and light sensitivity.

Patients have to be overall healthy without a history of skin cancer, keloidal scarring, localized or active infection, immunodeficiency disorders, and light sensitivity. Per PI discretion, any serious medical condition that may interfere with the study. In addition, patients who have been taking isotretinoin for a period of 6 months before treatment will be excluded.

Patients will have photographs taken at every visit prior to the laser treatments at week 0, week 4, and week 8. Photographs will also be taken at the week 24 follow-up visit. Photos will then be assessed by qualified blinded reviewers for comparison.

ELIGIBILITY:
Inclusion Criteria:

* Men and women with Fitzpatrick skin types I through V and facial acne scarring of grades III-IV (moderate to severe) will be enrolled. Both sides of the participants' face should have similar amount and severity of acne scarring. Participants will be over 18 years old. Patients have to be otherwise healthy without a history of skin cancer, keloidal scarring, localized or active infection, immunodeficiency disorders, and light sensitivity.

Exclusion Criteria:

* Patients have to be overall healthy without a history of skin cancer, keloidal scarring, localized or active infection, immunodeficiency disorders, and light sensitivity. Per PI discretion, any serious medical condition that may interfere with the study. In addition, patients who have been taking isotretinoin for a period of 6 months before treatment will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-03-08 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David R Smart, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah MidValley Dermatology, Murray, Utah, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: half faces of subjects
Groups:
- 1,550 Laser: All subjects on this arm will be treated on this split-faced. This arm is looking at the side of the face treated with the 1,550-nanometer Fracionated Photothermolysis laser.
  1,550 fracionated photothermolysis laser vs. 755 picosecond laser: All subjects will have one side of their face treated with one laser, and the other side with the other laser.
- 755 Laser: All subjects on this arm will be treated on this split-faced. This arm is the side of their face will be treated with the 755-nanometer alexandrite picosecond laser.
  1,550 fracionated photothermolysis laser vs. 755 picosecond laser: All subjects will have one side of their face treated with one laser, and the other side with the other laser.
Period: Overall Study
Arm/Group | 1,550 Laser | 755 Laser
Started | 22; 22 half faces of subjects | 22; 22 half faces of subjects
Completed | 22; 22 half faces of subjects | 22; 22 half faces of subjects
Not Completed | 0; 0 half faces of subjects | 0; 0 half faces of subjects

BASELINE CHARACTERISTICS:
Population: There were 22 participants total, but each participate received each treatment on half of their face. Therefore, there are 22 participants in each arm, with at total of 22 participants. But there are 44 half faces analyzed in the trial.
Units Other Than Participants: half faces
Groups:
- 1,550 Laser: All subjects on this arm will be treated on this split-faced. This arm consists of the half-faces treated with the 1,550-nanometer Fracionated Photothermolysis laser.
  1,550 fracionated photothermolysis laser vs. 755 picosecond laser: All subjects will have one side of their face treated with one laser, and the other side with the other laser.
- 755 Laser: All subjects on this arm will be treated on this split-faced. This arm consists of the half-faces treated with the 755-nanometer alexandrite picosecond laser.
  1,550 fracionated photothermolysis laser vs. 755 picosecond laser: All subjects will have one side of their face treated with one laser, and the other side with the other laser.
- Total: Total of all reporting groups
Arm/Group | 1,550 Laser | 755 Laser | Total
Number analyzed (Participants) | 22 | 22 | 22
Number analyzed (half faces) | 22 | 22 | 44
Age, Categorical [Count of Participants; unit: Participants] — Population: Number of units analyzed was 2 per participant.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 22 | 22 | 44
    >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: the number of units analyzed was 2 per participant.
  years | 33 (14.28) | 33 (14.28) | 33 (14.28)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: the number of units analyzed was 2 per participant.
  Participants
    Female | 10 | 10 | 20
    Male | 12 | 12 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants] — Each participant received both lasers (one on each side of the face). So there are 22 participants total, however, there are 22 halves of faces on each treatment arm. Population: the number of units analyzed was 2 per participant.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 2 | 2 | 4
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 2 | 2 | 4
    White | 15 | 15 | 30
    More than one race | 3 | 3 | 6
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — Population: the number of units analyzed was 2 per participant.
  participants
    United States | 22 | 22 | 22

OUTCOME MEASURES:

1. Primary Outcome: Number of Half Faces to Achieve at Least 25% Improvement in Acne Scarring at Week 24 by Blinded Photo Reviewer
Description: Change in Baseline acne scarring compared to week 24 measured by photographic review. Measured by blinded reviewer assessments of photographs.
Time Frame: Photos will be taken at week 0, week 4, week 8, and week 24.
Measure: Count of Units; unit: half faces
Units Other Than Participants: half faces
Arm/Group | 1,550 Laser | 755 Laser
Number analyzed (Participants) | 22 | 22
Number analyzed (half faces) | 22 | 22
half faces | 18 | 17

ADVERSE EVENTS:
Time Frame: Adverse events (anticipated and unanticipated) related to study treatments/procedures (based on the judgment of an investigator) were collected from the time of signed consent through week 24.
Description: The adverse events collected for this study differ from the clinicaltrials.gov definition in that the adverse events collected were only considered related to the participant's participation in the research.
Arm/Group | 1,550 Laser | 755 Laser
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 22/22 | 22/22
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1,550 Laser (N=22) | 755 Laser (N=22)
Transient Erythema (Skin and subcutaneous tissue disorders) | 22 (22) | 22 (22)
Transient Crusting or Blistering (Skin and subcutaneous tissue disorders) | 22 (22) | 22 (22)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-01): https://cdn.clinicaltrials.gov/large-docs/49/NCT03988049/Prot_SAP_000.pdf